CLINICAL TRIAL: NCT01199861
Title: A 3-month Blinded, Randomized, Multicenter, Placebo-controlled Study to Evaluate the Effect of Treatment With Fingolimod on the Immune Response Following Seasonal Influenza Vaccination and Tetanus Toxoid Booster Injection in Patients With Relapsing Forms of Multiple Sclerosis (MS)
Brief Title: Effect of Treatment With Fingolimod on the Immune Response Following Seasonal Flu Vaccination and Tetanus Booster Injection in Patients With Relapsing Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFTY720D2320; 2010-019028-30 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-05

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing multiple sclerosis; MS; Immune response
MeSH Terms: interventions — Fingolimod Hydrochloride; Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Fingolimod (Experimental): Participants received Fingolimod 0.5 mg capsules orally once daily for 12 weeks. At Week 6 of study treatment participants received a seasonal influenza vaccination and a tetanus booster vaccination.
  Interventions: Drug: Fingolimod; Biological: Seasonal influenza vaccine; Biological: Tetanus toxoid vaccine
- Placebo (Placebo Comparator): Participants received placebo tablets orally once daily for 12 weeks. At Week 6 of study treatment participants received a seasonal influenza vaccination and a tetanus booster vaccination.
  Interventions: Drug: Placebo; Biological: Seasonal influenza vaccine; Biological: Tetanus toxoid vaccine

INTERVENTIONS:
Drug: Fingolimod — Fingolimod 0.5 mg capsules for oral administration.
  Other Names: FTY720
  Arms: Fingolimod
Drug: Placebo — Matching placebo capsules for oral administration.
  Arms: Placebo
Biological: Seasonal influenza vaccine — Commercially available injectable influenza vaccine for the 2010/11 influenza season.
  Other Names: Agrippal (TM)
Biological: Tetanus toxoid vaccine — Commercially available tetanus toxoid vaccine booster injection.
  Other Names: Tetanol (TM)

SUMMARY:
This study will evaluate the effect of treatment with fingolimod on the immune response following seasonal influenza vaccination and tetanus booster injection in patients with relapsing MS.

ELIGIBILITY:
Inclusion Criteria:

* Must have relapsing MS
* Must have lifetime tetanus vaccination
* Agree to receive 2010/2011 seasonal influenza vaccine and tetanus toxoid booster injection

Exclusion Criteria:

* Patients with a type of MS that is not relapsing
* Patients with history of chronic immune disease
* Certain cancers
* Diabetic patients with certain eye disorders
* Patients who are on certain immunosuppressive medications or heart medications
* Patients with certain heart conditions
* Patients with certain lung conditions
* Patients who have already received the 2010/2011 seasonal influenza vaccine

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Belgium (5):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
- Canada (3):
  - Novartis Investigative Site, Nepean, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke
- Finland (2):
  - Novartis Investigative Site, Seinäjoki
  - Novartis Investigative Site, Turku
- France (4):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Guatemala City, Guatemala
- Poland (2):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
- Spain (3):
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigational Site, Basel, Switzerland
- United Kingdom (2):
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 2:1 ratio to fingolimod 0.5 mg once daily or matching placebo.
Period: Overall Study
Arm/Group | Fingolimod | Placebo
Started | 95 | 43
Completed | 93 | 43
Not Completed | 2 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Placebo | Total
Number analyzed (Participants) | 95 | 43 | 138
Age Continuous [Mean (Standard Deviation); unit: years] | 37.4 (8.37) | 39.2 (8.67) | 37.9 (8.48)
Age, Customized [Number; unit: participants]
  18-30 | 25 | 8 | 33
  31-40 | 35 | 14 | 49
  41-55 | 35 | 21 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 29 | 94
  Male | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Immune Response 3 Weeks After Seasonal Influenza Vaccination
Description: Percentage of participants who responded to treatment with the seasonal influenza vaccine 3 weeks after vaccination. Response was defined as patients fulfilling one of the following criteria for at least one of the three strains contained in the seasonal influenza vaccine:
  * Seroconversion: The pre-vaccination antibody titer measurement was <1:10 and the post-vaccination measurement is ≥1:40.
  * Significant increase in antibody titer: The pre-vaccination antibody titer measurement was ≥1:10 and the increase in antibody titer from this to the post-vaccination measurement is ≥ 4-fold.
Time Frame: Week 6 (pre-vaccination) and 3 weeks after vaccination (Study week 9)
Population: The full analysis set which includes all patients who were randomized and received at least 1 dose of study drug, and for whom data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 90 | 43
percentage of participants | 53.3 | 83.7

2. Secondary Outcome: Immune Response 6 Weeks After Seasonal Influenza Vaccination
Description: Percentage of participants who responded to treatment with the seasonal influenza vaccine 6 weeks after vaccination. Response was defined as patients fulfilling one of the following criteria for at least one of the three strains contained in the seasonal influenza vaccine:
  * Seroconversion: The pre-vaccination antibody titer measurement was <1:10 and the post-vaccination measurement is ≥1:40.
  * Significant increase in antibody titer: The pre-vaccination antibody titer measurement was ≥1:10 and the increase in antibody titer from this to the post-vaccination measurement is ≥ 4-fold.
Time Frame: Week 6 (pre-vaccination) and 6 weeks after vaccination (Study week 12).
Population: Full analysis set for whom data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 88 | 43
percentage of participants | 43.2 | 74.4

3. Secondary Outcome: Immune Response 3 Weeks After Tetanus Toxoid Booster
Description: Percentage of participants with an immune response to a single dose of tetanus toxoid three weeks after vaccination. A patient was considered a responder to tetanus toxoid booster vaccination if one of the following criteria was met:
  1. Seroconversion: The pre-vaccination antibody titer measurement was <0.1 IU/ml and the post-vaccination measurement was ≥0.4 IU/ml.
  2. Significant increase: The pre-vaccination antibody titer measurement was ≥0.1 IU/ml and the increase in antibody titer from this to the post-vaccination measurement was ≥4- fold.
Time Frame: Week 6 (pre-vaccination) and 3 weeks after vaccination (Study Week 9)
Population: Full analysis set for whom data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 90 | 43
percentage of participants | 40.0 | 60.5

4. Secondary Outcome: Immune Response 6 Weeks After Tetanus Toxoid Booster
Description: Percentage of participants with an immune response to a single dose of tetanus toxoid six weeks after vaccination. A patient was considered a responder to tetanus toxoid booster vaccination if one of the following criteria was met:
  1. Seroconversion: The pre-vaccination antibody titer measurement was <0.1 IU/ml and the post-vaccination measurement was ≥0.4 IU/ml.
  2. Significant increase: The pre-vaccination antibody titer measurement was ≥0.1 IU/ml and the increase in antibody titer from this to the post-vaccination measurement was ≥4- fold.
Time Frame: Week 6 (pre-vaccination) and 6 weeks after vaccination (Study Week 12)
Population: Full analysis set for whom data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 88 | 43
percentage of participants | 37.5 | 48.8

5. Secondary Outcome: Change From Baseline in Seasonal Influenza Vaccine Antibody-titer 3 Weeks After Vaccination
Description: Change from Baseline was expressed by the ratio of post-vaccination to pre-vaccination antibody titer for each of the three strains included in the seasonal influenza vaccine. Inhibition of an immune response to each strain included in the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo three weeks after a single dose of seasonal influenza vaccine.
Time Frame: Pre-vaccination (Week 6) and 3 weeks after vaccination (Study Week 9).
Population: Full analysis set for whom data were available.
Measure: Number; unit: ratio
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 90 | 43
ratio
  A/California/7/09(H1N1) | 2.45 | 4.14
  A/Perth/16/2009(H3N2) | 0.49 | 0.36
  B/Brisbane/60/2008 | 1.34 | 2.40
Statistical Analysis 1: Comparison: Fingolimod vs Placebo; The inhibition of an immune response to the A/California/7/09 (H1N1) strain of the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo three weeks after a single dose of seasonal influenza vaccine; Test type: Superiority or Other; Percent Inhibition = 41.0 — One minus the back-transformed estimate for the treatment difference was interpreted as the relative inhibition of an immune response caused by fingolimod 0.5 mg compared to placebo; it was presented as a percentage and referred to as 'inhibition'
Statistical Analysis 2: Comparison: Fingolimod vs Placebo; The inhibition of an immune response to the A/Perth/16/2009 (H3N2) strain of the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo three weeks after a single dose of seasonal influenza vaccine; Test type: Superiority or Other; Percent Inhibition = -35.0 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Fingolimod vs Placebo; The inhibition of an immune response to the B/Brisbane/60/2008 strain of the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo three weeks after a single dose of seasonal influenza vaccine; Test type: Superiority or Other; Percent Inhibition = 44.0 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Seasonal Influenza Vaccine Antibody-titer 6 Weeks After Vaccination
Description: Change from Baseline was expressed by the ratio of post-vaccination to pre-vaccination antibody titer for each of the three strains included in the seasonal influenza vaccine. Inhibition of an immune response to each strain included in the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo six weeks after a single dose of seasonal influenza vaccine.
Time Frame: Pre-vaccination (Week 6) and 6 weeks after vaccination (Study Week 12).
Population: Full analysis set for whom data were available.
Measure: Number; unit: ratio
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 88 | 43
ratio
  A/California/7/09(H1N1) | 1.81 | 2.91
  A/Perth/16/2009(H3N2) | 0.36 | 0.28
  B/Brisbane/60/2008 | 1.08 | 2.07
Statistical Analysis 1: Comparison: Fingolimod vs Placebo; The inhibition of an immune response to the A/California/7/09 (H1N1) strain of the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo six weeks after a single dose of seasonal influenza vaccine; Test type: Superiority or Other; Percent Inhibition = 38.0 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Fingolimod vs Placebo; The inhibition of an immune response to the A/Perth/16/2009 (H3N2) strain of the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo six weeks after a single dose of seasonal influenza vaccine; Test type: Superiority or Other; Percent Inhibition = -28.0 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Fingolimod vs Placebo; The inhibition of an immune response to the B/Brisbane/60/2008 strain of the seasonal influenza vaccine was assessed by the relative difference of the geometric mean antibody titer ratio on fingolimod as compared to placebo six weeks after a single dose of seasonal influenza vaccine; Test type: Superiority or Other; Percent Inhibition = 48.0 — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Relationship to study drug was determined by the investigator (suspected/not suspected).
  A serious AE is defined as an event which fulfills one of the following criteria:
  * is fatal or life-threatening;
  * results in persistent or significant disability/incapacity;
  * constitutes a congenital anomaly/birth defect;
  * requires inpatient hospitalization or prolongation of existing hospitalization;
  * is medically significant, i.e., jeopardizes the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: From first dose of study drug until 45 days after the last dose of study drug (130 days).
Population: Safety set - all patients who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fingolimod | Placebo
Number analyzed (Participants) | 95 | 43
participants
  Any adverse event | 82 | 34
  AE related to study drug | 42 | 11
  Serious adverse event | 1 | 2
  Adverse events leading to discontinuation | 1 | 0

ADVERSE EVENTS:
Arm/Group | Fingolimod | Placebo
Serious Adverse Events (participants affected / at risk) | 1/95 | 2/43
Other Adverse Events (participants affected / at risk) | 51/95 | 22/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=95) | Placebo (N=43)
Herpes zoster (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=95) | Placebo (N=43)
Lymphopenia (Blood and lymphatic system disorders) | 10 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 3 | 3
Nasopharyngitis (Infections and infestations) | 15 | 8
Upper respiratory tract infection (Infections and infestations) | 11 | 6
Urinary tract infection (Infections and infestations) | 5 | 2
Headache (Nervous system disorders) | 18 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.